CLINICAL TRIAL: NCT00646945
Title: International, Randomized, Controled, Double-Blind Study Assessing Efficacy of Kalinox® 170 Bar During the Realization of Invasive Gestures in Adult Oncology
Brief Title: Study of the Efficacy of Kalinox® 170 Bar in Adult Oncology
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Air Liquide Santé International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 2006-003226-29
Record Dates: First submitted 2008-03-20; First posted 2008-03-31 (Estimated); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Cancer; Pain
Keywords: Patient in a oncology unit who has to undergo a painful or invasive procedure
MeSH Terms: conditions — Neoplasms; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): 50% Oxygen/50% Nitrous oxide premix (Kalinox 170 bar)
  Interventions: Drug: 50% Oxygen/50% Nitrous oxide premix (Kalinox 170 bar)
- B (Placebo Comparator): 50% oxygen/50% Nitrogen premix
  Interventions: Drug: 50% Oxygen/50% Nitrogen premix

INTERVENTIONS:
Drug: 50% Oxygen/50% Nitrous oxide premix (Kalinox 170 bar) — gas flow between 4 to 15 L/min
  Arms: A
Drug: 50% Oxygen/50% Nitrogen premix — gas flow between 4 to 15 L/min
  Arms: B

SUMMARY:
In the oncology practice, The National Union of the Centres of Fight Against the Cancer recently published the Standards, Options and Recommendations for the coverage of the pains provoked during the invasive gestures of a short duration realized at patients affected by cancer. These support the use of the Kalinox ® 170 bar as therapeutic alternative for the preparation of the painful procedures of a short duration such as spinal taps or osseous at the adult.The objective of this study thus is to clarify the appropriate efficiency and the tolerance of the equimolar mixture protoxide of nitrogen / oxygen during invasive procedures realized in adult oncology with regard to the analgesic reference methods and to the effect placebo leads by the accompaniment of the patient during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 year
* OMS between 0 to 3
* Patient who has to undergo an invasive gesture or a painful care
* Absence of contra-indication to the administration of the product

Exclusion Criteria:

* Patient already included in another incompatible study with this protocol
* Patient incapable of self-assessment by the EVA
* Confusional syndrome
* OMS > 3
* Patient already included in this protocol
* Exclusion criteria linked to the product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2007-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
pain measurement with visual analogue scale | EVA

SECONDARY OUTCOMES:
feasibility of the kalinox 170 bar in invasives gestures in oncology | opinion of the patent and the caregiver
surveillance of the appearance of secondary effects | examination by the investigator

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Alexis Vautrin, Vandœuvre-lès-Nancy, France

REFERENCES:
- [Result] Prise en charge de la douleur au cours des procédures invasives en cancérologie : efficacité et acceptabilité du mélange inhalé 50 % N2O/O2 (MEOPA) Pain management during invasive procedures in oncology: inhaled 50% N2O/O2 premix, an effective and well tolerated method I. Krakowski · D Baylot · G. Chvetzoff · E. Collin · R. Coulouma · F. Dixmerias · L. Feuvret · C. Freyssinet-Durand · E. Lauwers-Allot · D. Lossignol · C. Billoët Douleur analg. (2010) 23:113-120 DOI 10.1007/s11724-010-0197-5
- See also: Related Info — https://link.springer.com/article/10.1007/s11724-010-0197-5